CLINICAL TRIAL: NCT03527641
Title: Unidos Por la Salud/United for Health: Innovative Community-Academic Partnership for Type 2 Diabetes Prevention
Brief Title: United for Health: Type 2 Diabetes Prevention in Latino Teens
Acronym: UNITED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-6568
Record Dates: First submitted 2018-04-23; First posted 2018-05-17 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Prediabetic State; Insulin Resistance; Type2 Diabetes; Stress; Adolescent Development; Family Research
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Exercise; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more group conditions in parallel for the duration of the study - (1) Salud sin Barreras or (2) La Vida Saludable. Both of these programs meet for 6 weeks, twice per week for 12 total 2-hour sessions. Youth are assessed at baseline, post-treatment, and 6-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salud sin Barreras, Health without Barriers (Experimental): Salud sin Barreras is a manualized community-delivered program tailored for Latino families and their adolescent children at-risk for type 2 diabetes. Salud sin Barreras is based upon a lifestyle intervention called the Healthy Living Program (HeLP), which includes 6 weekly 2-hour nutrition/cooking sessions and 6 weekly 2-hour Multidisciplinary Sessions that include parent education on nutrition, fitness, goal-setting, parenting, and a brief mindfulness curriculum, a teen group physical fitness class, and a teen mindfulness curriculum called Learning 2 BREATHe. In between sessions, participants are encouraged to practice brief mindfulness skills in their daily lives and to complete the "homework" assignments, such as an audio-guided body scan. Participants have access to home-practice audio-recordings and will be queried about their completion of home-practice assignments.
  Interventions: Behavioral: CookingMatters; Behavioral: Parent Education; Behavioral: Physical Activity; Behavioral: Mindfulness-based Stress Reduction; Behavioral: Brief Mindfulness Intervention
- La Vida Saludable, Healthy Living (Active Comparator): The Health Living Program (HeLP) is a manualized community-delivered program tailored specifically for Latino families and children at-risk for adult obesity. HeLP includes 6 weekly 2-hour nutrition/cooking sessions and 6 weekly 2-hour Multidisciplinary Sessions, that include parent education on nutrition, fitness, goal-setting, and parenting, a teen group physical fitness class, and a teen health knowledge curriculum derived from a health education curriculum called Hey DURHAM.
  Interventions: Behavioral: CookingMatters; Behavioral: Parent Education; Behavioral: Physical Activity; Behavioral: Health Education

INTERVENTIONS:
Behavioral: CookingMatters — Nutrition education and hands-on cooking lessons for the whole family
Behavioral: Parent Education — Parenting, physical activity and nutrition education, and family health education for parents
Behavioral: Physical Activity — Physical fitness activities for teens
Behavioral: Health Education — Health knowledge curriculum for adolescents
  Other Names: Hey Durham
  Arms: La Vida Saludable, Healthy Living
Behavioral: Mindfulness-based Stress Reduction — Adolescent mindfulness curriculum
  Other Names: Learning to Breathe
  Arms: Salud sin Barreras, Health without Barriers
Behavioral: Brief Mindfulness Intervention — Parent-based education and experiential learning of mindfulness-based tools
  Other Names: Learning to Breathe, Parent Education
  Arms: Salud sin Barreras, Health without Barriers

SUMMARY:
This study pilots the feasibility and acceptability of a family-based lifestyle intervention for decreasing diabetes risk called "Salud sin Barreras" (meaning, "Health without Barriers") delivered in the community to Latino teens at risk for type 2 diabetes. This program combines traditional lifestyle intervention to change eating and physical activity with learning mindfulness-based stress reduction tools. We also are exploring how Salud sin Barreras lowers stress and improves insulin resistance in Latino teens, as compared to lifestyle-only intervention, the "La Vida Saludable" (meaning, the Healthy Living Program; HeLP).

DETAILED DESCRIPTION:
This study is a comparative effectiveness pilot trial to evaluate the feasibility and acceptability of a 12-session community-delivered, family-based type 2 diabetes preventative lifestyle intervention, delivered over 6 weeks, that includes mindfulness-based stress reduction training - "Salud sin Barreras" (meaning, "Health without Barriers") - in up to 50 Hispanic/Latino adolescents who are at-risk for developing type 2 diabetes. We also will estimate the effectiveness of Salud sin Barreras for lowering perceived stress and improving insulin resistance as compared to a time-matched lifestyle-only intervention, the "La Vida Saludable" (meaning, the Healthy Living Program; HeLP) in Hispanic/Latino adolescents at-risk for type 2 diabetes. In addition, we will estimate the impact of the Salud sin Barreras program, relative to HeLP, on the secondary outcomes of mindfulness, depressive symptoms, disinhibited eating behavior, sleep quality, physical activity, cortisol, and perceived impact of discrimination.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-15 years
* Identify as Hispanic/Latino
* English speaking
* At-risk for T2D by virtue of current BMI ≥ 85th percentile for age and sex by CDC 2000 standards and ≥ 1 first or second degree biological relative with T2D, prediabetes, or gestational diabetes
* Currently a Salud Family Health Center patient or willing to become a patient of Salud Family Health Center (required to complete medical assessments at Salud)

Exclusion Criteria:

* Major medical problem, including type 1 diabetes or T2D
* Reported psychiatric disorder that would impede compliance in the opinion of the investigators
* Started use of medication affecting mood or body weight, such as stimulants or anti-depressants within the past 3 months
* Any medical issues that could be acutely worsened by exercise such as severe or uncontrolled asthma or musculoskeletal problems
* Self-reported pregnancy in girls

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment/Enrollment | Up to 12 week period preceding the start of the intervention
  Feasibility of recruitment/enrollment for community-based family lifestyle intervention for Latino teens at-risk for type 2 diabetes as measured by number of qualifying participants following screening
Treatment Acceptability Questionnaire | 6 weeks
  Survey adapted from the Treatment Acceptability Questionnaire to assess acceptability and satisfaction with program participation; items are rated on a scale ranging from 1-5 with higher scores reflecting more positive acceptability
Perceived Stress Scale | 6 months
  Survey assessing perceptions of stress; the total score, calculated as the sum of all items, ranges from 0 to 60, with higher values reflecting more perceived stress
Homeostasis model assessment of insulin resistance (HOMA-IR) | 6 months
  Poor sensitivity of insulin to respond to and regulate glucose (blood sugar) as estimated from fasting glucose and insulin values

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale | 6 months
  Survey assessing propensity for present-moment attention; a total score is calculated as the sum of all items with a possible range of 15-90, with higher scores reflecting greater mindfulness (positive outcome) and lower scores, less mindfulness (worse outcome)
Center for Epidemiologic Studies-Depression Scale | 6 months
  Survey measure of symptoms of depression; a total score is calculated as the sum of all items with a possible range of 0-60, with higher scores reflecting more depressive symptoms
Emotional Eating Scale Adapted for Children and Adolescents | 6 months
  Survey measure of eating in response to negative emotions; subscales include eating in response to depression, eating in response to anger/anxiety/frustration, and eating in response to boredom with subscales calculated as the average of items; subscales range from 1-5 with higher scores indicating more emotional eating
Actigraph GT3x Sleep Time | 6 months
  Total sleep time as assessed by wrist-worn accelerometry
Actigraph GT3x Physical Activity | 6 months
  Total amount of minutes spent in light, moderate, and vigorous activity as assessed by wrist-worn accelerometry
Cortisol | 6 weeks
  Stress hormone as assessed by salivary swab
Everyday Discrimination Scale | 6 months
  Survey assessing perceived impact of discrimination; a total score is calculated from the sum of all items, with the total score ranging from 1 to 54, with higher scores indicating higher levels of perceived discrimination

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Salud Family Health Center, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No